CLINICAL TRIAL: NCT00408876
Title: Protocol F1J-MC-HMEO Duloxetine Versus Placebo in the Treatment of Chronic Low Back Pain
Brief Title: Duloxetine Versus Placebo in Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10545; F1J-MC-HMEO
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-11

CONDITIONS: Back Pain Without Radiation
MeSH Terms: conditions — Back Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Duloxetine 20 mg (Experimental): duloxetine 20 mg once a day (QD), by mouth (PO) for 13 weeks
  Interventions: Drug: Duloxetine
- Duloxetine 60 mg (Experimental): duloxetine 30 mg once a day (QD), by mouth (PO) for 1 week then duloxetine 60 mg QD, PO for 12 weeks
  Interventions: Drug: Duloxetine
- Duloxetine 120 mg (Experimental): duloxetine 30 mg once a day (QD), by mouth (PO) for 1 week followed by duloxetine 60 mg QD, PO for 1 week, then duloxetine 120 mg QD, PO for 11 weeks
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): placebo once a day (QD), by mouth (PO) for 13 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 120 mg; Duloxetine 20 mg; Duloxetine 60 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of your participation in this study is to help answer the following research question, and not to provide you treatment for your condition--Whether duloxetine once daily can help patients with Chronic Low Back Pain.

ELIGIBILITY:
Inclusion Criteria: - Male/Female outpatients 18 years of age with chronic low back pain. Exclusion Criteria: - You have a serious or unstable disease of the heart or blood vessels, liver, kidney, lungs, or blood-related illness, problems with decreased blood flow to arms and legs (peripheral vascular disease), or other medical conditions, or psychiatric conditions that, in the opinion of the investigator, would affect your participation or be likely to lead to hospitalization during the course of the study. - Have acute liver injury (such as hepatitis) or severe cirrhosis. - Have had previous exposure to duloxetine. - Have a body mass index (BMI) over 40. - Have major depressive disorder. - Require daily narcotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Tampa, Florida

REFERENCES:
- [Derived] Williamson OD, Schroer M, Ruff DD, Ahl J, Margherita A, Sagman D, Wohlreich MM. Onset of response with duloxetine treatment in patients with osteoarthritis knee pain and chronic low back pain: a post hoc analysis of placebo-controlled trials. Clin Ther. 2014 Apr 1;36(4):544-51. doi: 10.1016/j.clinthera.2014.02.009. Epub 2014 Mar 17. PMID 24650448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Started | 59 | 116 | 112 | 117
Completed | 43 | 80 | 62 | 82
Not Completed | 16 | 36 | 50 | 35
Not completed — Adverse Event | 9 | 17 | 27 | 10
Not completed — Withdrawal by Subject | 3 | 6 | 6 | 14
Not completed — Lack of Efficacy | 2 | 4 | 5 | 6
Not completed — Lost to Follow-up | 1 | 6 | 5 | 2
Not completed — Protocol Violation | 0 | 3 | 4 | 3
Not completed — Physician Decision | 1 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo | Total
Number analyzed (Participants) | 59 | 116 | 112 | 117 | 404
Age Continuous [Mean (Standard Deviation); unit: years] | 52.93 (12.81) | 53.32 (14.69) | 54.92 (14.77) | 53.97 (13.52) | 53.89 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 67 | 65 | 64 | 232
  Male | 23 | 49 | 47 | 53 | 172
Region of Enrollment [Number; unit: participants]
  United States | 46 | 92 | 85 | 93 | 316
  Argentina | 13 | 24 | 27 | 24 | 88
Race/Ethnicity [Number; unit: participants]
  African | 7 | 11 | 5 | 10 | 33
  Caucasian | 46 | 91 | 92 | 93 | 322
  East Asian | 0 | 1 | 1 | 1 | 3
  Hispanic | 6 | 13 | 11 | 11 | 41
  West Asian | 0 | 0 | 3 | 1 | 4
  Native American | 0 | 0 | 0 | 1 | 1
Beck Depression Inventory-II Total Score [Mean (Standard Deviation); unit: units on a scale] — A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
  units on a scale | 6.02 (6.33) | 7.05 (7.17) | 5.20 (5.00) | 6.15 (7.52) | 6.12 (6.64)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 30.42 (4.54) | 28.85 (4.73) | 29.23 (4.68) | 28.67 (4.89) | 29.13 (4.75)
Brief Pain Inventory (BPI) 24-Hour Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 6.34 (1.64) | 5.93 (1.67) | 6.04 (1.63) | 6.14 (1.66) | 6.08 (1.65)
Clinical Global Impressions of Severity (CGI-S) Scale [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.05 (1.41) | 3.54 (1.40) | 3.58 (1.33) | 3.66 (1.30) | 3.66 (1.36)
Duration of Chronic Low Back Pain [Mean (Standard Deviation); unit: years] | 12.50 (11.65) | 10.48 (11.07) | 13.94 (12.97) | 10.29 (9.53) | 11.68 (11.38)
Patient Global Impressions of Severity (PGI-S) Scale [Mean (Standard Deviation); unit: units on a scale] — Measures patient's perception of severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (extremely ill ).
  units on a scale | 2.78 (1.69) | 2.63 (1.78) | 2.25 (1.58) | 2.38 (1.60) | 2.48 (1.67)
Roland-Morris Disability Questionnaire Total Score [Mean (Standard Deviation); unit: units on a scale] — Roland-Morris questionnaire was completed by the patient and measured the degree of disability due to back pain. The questionnaire consists of 24 statements and the patient was instructed to put a mark next to each appropriate statement. The number of statements marked was added up by the clinician and a total score was given. The total score ranges from 0 (no disability) to 24 (severe disability).
  units on a scale | 10.00 (4.82) | 8.91 (4.56) | 8.72 (4.82) | 8.32 (4.92) | 8.85 (4.79)
Weekly Mean of 24-Hour Average Pain Severity [Mean (Standard Deviation); unit: units on a scale] — 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean, with scores ranging from 0 (no pain) to 10 (worst possible pain).
  units on a scale | 6.42 (1.39) | 6.18 (1.44) | 6.06 (1.45) | 6.18 (1.25) | 6.18 (1.38)
Weekly Mean of 24-Hour Worst Pain Severity [Mean (Standard Deviation); unit: units on a scale] — 24-hour worst pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean, with scores ranging from 0 (no pain) to 10 (worst possible pain).
  units on a scale | 7.41 (1.31) | 7.22 (1.32) | 7.22 (1.27) | 7.35 (1.20) | 7.29 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 1 in Weekly Mean of the 24-hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 1), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 1
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 104 | 108 | 110
units on a scale | -0.54 (0.18) | -0.53 (0.13) | -0.71 (0.13) | -0.39 (0.13)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.503, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.447, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.084, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.964, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.451, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.333, Repeated Measures

2. Secondary Outcome: Patient's Global Impression - Improvement (PGI-I) at Week 13 Endpoint
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from
  1 (very much better) to 7 (very much worse).
Time Frame: Week 13
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value. Endpoint is the last non-missing measure from Week 4 to Week 13. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 57 | 108 | 107 | 114
units on a scale | 2.72 (0.17) | 2.44 (0.13) | 2.66 (0.13) | 2.93 (0.13)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.318, t-test, 2 sided; Mean Difference (Net) = -0.21, 95% CI [-0.62 to 0.20]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.005, t-test, 2 sided; Mean Difference (Net) = -0.49, 95% CI [-0.83 to -0.15]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.124, t-test, 2 sided; Mean Difference (Net) = -0.27, 95% CI [-0.61 to 0.07]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.183, t-test, 2 sided; Mean Difference (Net) = -0.28, 95% CI [-0.70 to 0.13]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.778, t-test, 2 sided; Mean Difference (Net) = -0.06, 95% CI [-0.48 to 0.36]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.210, t-test, 2 sided; Mean Difference (Net) = 0.22, 95% CI [-0.13 to 0.57]

3. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Roland-Morris Disability Questionnaire (RMDQ) Total Score
Description: Roland-Morris questionnaire was completed by the patient and measured the degree of disability due to back pain. The questionnaire consists of 24 statements and the patient was instructed to put a mark next to each appropriate statement. The number of statements marked was added up by the clinician and a total score was given. The total score ranges from 0 (no disability) to 24 (severe disability).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 52 | 83 | 83 | 92
units on a scale | -2.29 (0.56) | -2.74 (0.44) | -2.88 (0.45) | -1.33 (0.43)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.161, t-test, 2 sided; Mean Difference (Net) = -0.97, 95% CI [-2.32 to 0.39]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.019, t-test, 2 sided; Mean Difference (Net) = -1.41, 95% CI [-2.59 to -0.24]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.010, t-test, 2 sided; Mean Difference (Net) = -1.56, 95% CI [-2.74 to -0.38]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.526, t-test, 2 sided; Mean Difference (Net) = -0.45, 95% CI [-1.83 to 0.94]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.397, t-test, 2 sided; Mean Difference (Net) = -0.59, 95% CI [-1.96 to 0.78]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.813, t-test, 2 sided; Mean Difference (Net) = -0.15, 95% CI [-1.35 to 1.06]

4. Secondary Outcome: Change From Baseline to Week 13 Endpoint in the 11-point Likert Scale, Weekly Mean 24-Hour Night Pain Score
Description: The 11-point Likert scale was used for assessment of 24-hour night pain and evaluated as weekly means. Scores range from from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 110 | 109 | 113
units on a scale | -1.77 (0.27) | -2.15 (0.20) | -2.47 (0.20) | -1.91 (0.19)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.657, t-test, 2 sided; Mean Difference (Net) = 0.15, 95% CI [-0.50 to 0.79]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.384, t-test, 2 sided; Mean Difference (Net) = -0.23, 95% CI [-0.76 to 0.29]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.040, t-test, 2 sided; Mean Difference (Net) = -0.56, 95% CI [-1.10 to -0.03]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.253, t-test, 2 sided; Mean Difference (Net) = -0.38, 95% CI [-1.03 to 0.27]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.034, t-test, 2 sided; Mean Difference (Net) = -0.71, 95% CI [-1.36 to -0.05]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.232, t-test, 2 sided; Mean Difference (Net) = -0.33, 95% CI [-0.86 to 0.21]

5. Secondary Outcome: Change From Baseline to Week 13 Endpoint in the 11-point Likert Scale, Weekly Mean of Worst Pain Score
Description: The 11-point Likert scale was used for assessment of 24-hour worst pain and evaluated as weekly means. Scores range from from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 110 | 109 | 113
units on a scale | -1.77 (0.30) | -2.46 (0.22) | -2.40 (0.22) | -2.10 (0.22)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.365, t-test, 2 sided; Mean Difference (Net) = 0.33, 95% CI [-0.39 to 1.05]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.232, t-test, 2 sided; Mean Difference (Net) = -0.36, 95% CI [-0.95 to 0.23]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.314, t-test, 2 sided; Mean Difference (Net) = -0.30, 95% CI [-0.90 to 0.29]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.062, t-test, 2 sided; Mean Difference (Net) = -0.69, 95% CI [-1.41 to 0.03]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.083, t-test, 2 sided; Mean Difference (Net) = -0.64, 95% CI [-1.36 to 0.08]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.859, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI [-0.54 to 0.65]

6. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Clinical Global Impression of Severity
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 108 | 107 | 112
units on a scale | -0.53 (0.14) | -0.94 (0.11) | -1.06 (0.11) | -0.53 (0.10)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.984, t-test, 2 sided; Mean Difference (Net) = 0.00, 95% CI [-0.34 to 0.34]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; Mean Difference (Net) = -0.41, 95% CI [-0.70 to -0.13]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -0.53, 95% CI [-0.81 to -0.24]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.018, t-test, 2 sided; Mean Difference (Net) = -0.42, 95% CI [-0.76 to -0.07]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Mean Difference (Net) = -0.53, 95% CI [-0.87 to -0.19]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.442, t-test, 2 sided; Mean Difference (Net) = -0.11, 95% CI [-0.40 to 0.17]

7. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Severity (BPI-S) - Worst Pain Score
Description: A self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 108 | 108 | 113
units on a scale | -1.78 (0.35) | -2.77 (0.25) | -2.78 (0.26) | -2.09 (0.25)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.464, t-test, 2 sided; Mean Difference (Net) = 0.31, 95% CI [-0.52 to 1.14]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.052, t-test, 2 sided; Mean Difference (Net) = -0.68, 95% CI [-1.36 to 0.00]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.052, t-test, 2 sided; Mean Difference (Net) = -0.68, 95% CI [-1.37 to 0.01]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.021, t-test, 2 sided; Mean Difference (Net) = -0.99, 95% CI [-1.83 to -0.15]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.020, t-test, 2 sided; Mean Difference (Net) = -0.99, 95% CI [-1.83 to -0.16]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.988, t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI [-0.70 to 0.69]

8. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Severity (BPI-S) - Least Pain Score
Description: A self-reported scale that measures the severity of pain based on the least pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 108 | 108 | 113
units on a scale | -1.30 (0.29) | -2.06 (0.21) | -2.16 (0.21) | -1.51 (0.20)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.543, t-test, 2 sided; Mean Difference (Net) = 0.21, 95% CI [-0.46 to 0.88]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.053, t-test, 2 sided; Mean Difference (Net) = -0.55, 95% CI [-1.10 to 0.01]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.024, t-test, 2 sided; Mean Difference (Net) = -0.65, 95% CI [-1.21 to -0.09]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.030, t-test, 2 sided; Mean Difference (Net) = -0.75, 95% CI [-1.43 to -0.07]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.014, t-test, 2 sided; Mean Difference (Net) = -0.85, 95% CI [-1.54 to -0.17]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.727, t-test, 2 sided; Mean Difference (Net) = -0.10, 95% CI [-0.66 to 0.46]

9. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Severity (BPI-S) - Average Pain Score
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 108 | 108 | 113
units on a scale | -1.79 (0.30) | -2.50 (0.22) | -2.45 (0.22) | -1.87 (0.22)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.813, t-test, 2 sided; Mean Difference (Net) = 0.09, 95% CI [-0.63 to 0.80]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.035, t-test, 2 sided; Mean Difference (Net) = -0.63, 95% CI [-1.21 to -0.04]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.054, t-test, 2 sided; Mean Difference (Net) = -0.58, 95% CI [-1.17 to 0.01]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.051, t-test, 2 sided; Mean Difference (Net) = -0.71, 95% CI [-1.43 to 0.00]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.070, t-test, 2 sided; Mean Difference (Net) = -0.67, 95% CI [-1.39 to 0.05]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.872, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI [-0.54 to 0.64]

10. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Severity (BPI-S) - Pain Right Now Score
Description: A self-reported scale that measures the severity of pain based on the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 108 | 108 | 113
units on a scale | -1.63 (0.33) | -2.67 (0.24) | -2.61 (0.24) | -1.74 (0.24)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.790, t-test, 2 sided; Mean Difference (Net) = 0.11, 95% CI [-0.68 to 0.89]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.005, t-test, 2 sided; Mean Difference (Net) = -0.93, 95% CI [-1.57 to -0.28]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Mean Difference (Net) = -0.87, 95% CI [-1.52 to -0.22]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.011, t-test, 2 sided; Mean Difference (Net) = -1.03, 95% CI [-1.83 to -0.24]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.016, t-test, 2 sided; Mean Difference (Net) = -0.97, 95% CI [-1.77 to -0.18]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.857, t-test, 2 sided; Mean Difference (Net) = 0.06, 95% CI [-0.60 to 0.72]

11. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - General Activity
Description: A self-reported scale that measures the interference of pain in the past 24 hours on general acitivity. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.99 (0.33) | -2.52 (0.24) | -2.36 (0.25) | -1.97 (0.24)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.948, t-test, 2 sided; Mean Difference (Net) = -0.03, 95% CI [-0.81 to 0.76]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.096, t-test, 2 sided; Mean Difference (Net) = -0.55, 95% CI [-1.20 to 0.10]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.239, t-test, 2 sided; Mean Difference (Net) = -0.39, 95% CI [-1.05 to 0.26]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.196, t-test, 2 sided; Mean Difference (Net) = -0.53, 95% CI [-1.32 to 0.27]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.367, t-test, 2 sided; Mean Difference (Net) = -0.37, 95% CI [-1.17 to 0.43]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.637, t-test, 2 sided; Mean Difference (Net) = 0.16, 95% CI [-0.50 to 0.82]

12. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Mood
Description: A self-reported scale that measures the interference of pain in the past 24 hours on mood. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.75 (0.30) | -2.52 (0.22) | -1.96 (0.22) | -1.70 (0.21)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.887, t-test, 2 sided; Mean Difference (Net) = -0.05, 95% CI [-0.76 to 0.65]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Mean Difference (Net) = -0.81, 95% CI [-1.40 to -0.23]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.392, t-test, 2 sided; Mean Difference (Net) = -0.26, 95% CI [-0.84 to 0.33]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.036, t-test, 2 sided; Mean Difference (Net) = -0.76, 95% CI [-1.48 to -0.05]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.573, t-test, 2 sided; Mean Difference (Net) = -0.20, 95% CI [-0.92 to 0.51]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.064, t-test, 2 sided; Mean Difference (Net) = 0.56, 95% CI [-0.03 to 1.15]

13. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Walking Ability
Description: A self-reported scale that measures the interference of pain in the past 24 hours on walking ability. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.79 (0.34) | -2.33 (0.25) | -1.89 (0.25) | -1.43 (0.24)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.374, t-test, 2 sided; Mean Difference (Net) = -0.36, 95% CI [-1.15 to 0.43]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.007, t-test, 2 sided; Mean Difference (Net) = -0.90, 95% CI [-1.55 to -0.25]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.169, t-test, 2 sided; Mean Difference (Net) = -0.46, 95% CI [-1.12 to 0.20]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.182, t-test, 2 sided; Mean Difference (Net) = -0.54, 95% CI [-1.35 to 0.26]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.802, t-test, 2 sided; Mean Difference (Net) = -0.10, 95% CI [-0.91 to 0.70]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.191, t-test, 2 sided; Mean Difference (Net) = 0.44, 95% CI [-0.22 to 1.11]

14. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Normal Work
Description: A self-reported scale that measures the interference of pain in the past 24 hours on normal work. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -2.20 (0.36) | -2.67 (0.26) | -2.38 (0.26) | -1.95 (0.26)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.556, t-test, 2 sided; Mean Difference (Net) = -0.25, 95% CI [-1.10 to 0.59]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.041, t-test, 2 sided; Mean Difference (Net) = -0.73, 95% CI [-1.42 to -0.03]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.220, t-test, 2 sided; Mean Difference (Net) = -0.44, 95% CI [-1.14 to 0.26]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.278, t-test, 2 sided; Mean Difference (Net) = -0.47, 95% CI [-1.33 to 0.38]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.673, t-test, 2 sided; Mean Difference (Net) = -0.18, 95% CI [-1.04 to 0.68]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.422, t-test, 2 sided; Mean Difference (Net) = 0.29, 95% CI [-0.42 to 1.00]

15. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Relations With Other People
Description: A self-reported scale that measures the interference of pain in the past 24 hours on relations with other people. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.33 (0.27) | -1.86 (0.20) | -1.27 (0.20) | -0.94 (0.19)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.234, t-test, 2 sided; Mean Difference (Net) = -0.39, 95% CI [-1.03 to 0.25]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -0.93, 95% CI [-1.46 to -0.40]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.213, t-test, 2 sided; Mean Difference (Net) = -0.34, 95% CI [-0.87 to 0.20]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.105, t-test, 2 sided; Mean Difference (Net) = -0.54, 95% CI [-1.19 to 0.11]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.876, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI [-0.60 to 0.70]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.033, t-test, 2 sided; Mean Difference (Net) = 0.59, 95% CI [0.05 to 1.13]

16. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Sleep
Description: A self-reported scale that measures the interference of pain in the past 24 hours on sleep. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.59 (0.32) | -2.48 (0.24) | -2.12 (0.24) | -1.63 (0.23)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.925, t-test, 2 sided; Mean Difference (Net) = 0.04, 95% CI [-0.73 to 0.80]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.008, t-test, 2 sided; Mean Difference (Net) = -0.85, 95% CI [-1.49 to -0.22]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.132, t-test, 2 sided; Mean Difference (Net) = -0.49, 95% CI [-1.12 to 0.15]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.024, t-test, 2 sided; Mean Difference (Net) = -0.89, 95% CI [-1.67 to -0.12]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.184, t-test, 2 sided; Mean Difference (Net) = -0.52, 95% CI [-1.30 to 0.25]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.262, t-test, 2 sided; Mean Difference (Net) = 0.37, 95% CI [-0.27 to 1.01]

17. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Enjoyment of Life
Description: A self-reported scale that measures the interference of pain in the past 24 hours on enjoyment of life. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.84 (0.32) | -2.49 (0.24) | -1.86 (0.24) | -1.76 (0.23)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.849, t-test, 2 sided; Mean Difference (Net) = -0.07, 95% CI [-0.84 to 0.69]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.024, t-test, 2 sided; Mean Difference (Net) = -0.73, 95% CI [-1.36 to -0.10]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.773, t-test, 2 sided; Mean Difference (Net) = -0.09, 95% CI [-0.73 to 0.54]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.097, t-test, 2 sided; Mean Difference (Net) = -0.66, 95% CI [-1.43 to 0.12]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.960, t-test, 2 sided; Mean Difference (Net) = -0.02, 95% CI [-0.79 to 0.75]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.052, t-test, 2 sided; Mean Difference (Net) = 0.64, 95% CI [0.00 to 1.28]

18. Primary Outcome: Change From Baseline to Week 2 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 2), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 2
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 53 | 102 | 102 | 106
units on a scale | -0.84 (0.25) | -0.91 (0.18) | -1.22 (0.18) | -0.75 (0.17)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.756, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.507, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.056, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.816, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.208, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.212, Repeated Measures

19. Primary Outcome: Change From Baseline to Week 3 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 3), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 3
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 50 | 103 | 97 | 107
units on a scale | -1.05 (0.26) | -1.58 (0.18) | -1.71 (0.19) | -1.01 (0.18)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.885, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.026, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.007, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.095, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.040, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.635, Repeated Measures

20. Primary Outcome: Change From Baseline to Week 4 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 4), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 4
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 49 | 101 | 93 | 104
units on a scale | -1.20 (0.26) | -1.70 (0.18) | -2.17 (0.19) | -1.02 (0.18)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.575, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.009, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.115, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.002, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.072, Repeated Measures

21. Primary Outcome: Change From Baseline to Week 5 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 5), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 5
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 46 | 89 | 70 | 91
units on a scale | -1.45 (0.25) | -1.94 (0.18) | -2.25 (0.18) | -1.26 (0.18)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.516, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.006, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.112, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.010, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.219, Repeated Measures

22. Primary Outcome: Change From Baseline to Week 6 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 6), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 6
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 44 | 93 | 73 | 93
units on a scale | -1.64 (0.24) | -2.10 (0.17) | -2.28 (0.18) | -1.34 (0.17)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.309, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.001, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.116, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.033, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.480, Repeated Measures

23. Primary Outcome: Change From Baseline to Week 7 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 7), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 7
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 44 | 91 | 72 | 93
units on a scale | -1.68 (0.24) | -2.17 (0.17) | -2.36 (0.18) | -1.57 (0.17)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.709, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.012, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.097, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.023, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.435, Repeated Measures

24. Primary Outcome: Change From Baseline to Week 8 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 8), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 8
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 43 | 85 | 65 | 80
units on a scale | -1.68 (0.24) | -2.29 (0.17) | -2.49 (0.18) | -1.65 (0.17)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.931, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.007, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.036, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.007, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.416, Repeated Measures

25. Primary Outcome: Change From Baseline to Week 9 in Weekly Mean of the 24-Hour Average Pain Scores
Description: as for outcome 1
Time Frame: Baseline, Week 9
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 44 | 85 | 64 | 88
units on a scale | -1.57 (0.23) | -2.21 (0.17) | -2.45 (0.18) | -1.71 (0.16)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.634, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.031, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.002, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.026, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.003, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.313, Repeated Measures

26. Primary Outcome: Change From Baseline to Week 10 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 10), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 10
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 43 | 83 | 60 | 87
units on a scale | -1.77 (0.23) | -2.24 (0.17) | -2.58 (0.18) | -1.73 (0.16)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.910, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.026, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.090, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.006, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.171, Repeated Measures

27. Primary Outcome: Change From Baseline to Week 11 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 11), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 11
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 41 | 81 | 61 | 85
units on a scale | -1.88 (0.23) | -2.32 (0.17) | -2.62 (0.19) | -1.79 (0.16)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.733, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.022, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.128, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.013, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.225, Repeated Measures

28. Primary Outcome: Change From Baseline to Week 12 in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 12), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 12
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 39 | 78 | 57 | 80
units on a scale | -1.87 (0.24) | -2.34 (0.17) | -2.46 (0.19) | -1.91 (0.17)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.890, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.079, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.035, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.117, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.060, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.647, Repeated Measures

29. Primary Outcome: Change From Baseline to Week 13 Endpoint in Weekly Mean of the 24-Hour Average Pain Scores
Description: 24-hour average pain severity scores recorded daily on an 11-point Likert scale, evaluated as a weekly mean (Week 13), with scores ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 13
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 41 | 74 | 56 | 74
units on a scale | -1.74 (0.25) | -2.50 (0.18) | -2.42 (0.20) | -2.10 (0.18)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.243, Repeated Measures
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.110, Repeated Measures
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.236, Repeated Measures
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.014, Repeated Measures
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.036, Repeated Measures
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.756, Repeated Measures

30. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Brief Pain Inventory Interference (BPI-I) Score - Average Interference
Description: A self-reported scale that measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 108 | 113
units on a scale | -1.84 (0.26) | -2.40 (0.19) | -1.92 (0.19) | -1.61 (0.19)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.465, t-test, 2 sided; Mean Difference (Net) = -0.23, 95% CI [-0.84 to 0.39]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Net) = -0.79, 95% CI [-1.30 to -0.29]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.233, t-test, 2 sided; Mean Difference (Net) = -0.31, 95% CI [-0.82 to 0.20]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.075, t-test, 2 sided; Mean Difference (Net) = -0.56, 95% CI [-1.19 to 0.06]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.798, t-test, 2 sided; Mean Difference (Net) = -0.08, 95% CI [-0.71 to 0.54]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.066, t-test, 2 sided; Mean Difference (Net) = 0.48, 95% CI [-0.03 to 1.00]

31. Secondary Outcome: Response to Treatment, as Defined by a 30% Reduction of Weekly Mean Score in 24-hour Average Pain Severity Ratings, Last Observation Carried Forward
Time Frame: Baseline to Week 13
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 110 | 109 | 113
participants | 23 | 59 | 63 | 49
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.869, Fisher Exact
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.141, Fisher Exact
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.033, Fisher Exact
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.142, Fisher Exact
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.049, Fisher Exact
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.587, Fisher Exact

32. Secondary Outcome: Response to Treatment, as Defined by a 50% Reduction of Weekly Mean Score in 24-hour Average Pain Severity Ratings, Last Observation Carried Forward
Time Frame: Baseline to Week 13
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 110 | 109 | 113
participants | 12 | 38 | 40 | 33
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.356, Fisher Exact
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.472, Fisher Exact
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.255, Fisher Exact
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.107, Fisher Exact
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.053, Fisher Exact
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.779, Fisher Exact

33. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Athens Insomnia Scale
Description: Estimates sleep difficulty. Consists of 8 items rated on a 4-point scale of 0 (no problem at all) to 3 (very serious problem). Total score of the 8-item version ranges from 0-24.
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 101 | 99 | 107
units on a scale | -1.43 (0.53) | -2.30 (0.39) | -0.93 (0.40) | -1.23 (0.38)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.747, t-test, 2 sided; Mean Difference (Net) = -0.21, 95% CI [-1.47 to 1.06]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.045, t-test, 2 sided; Mean Difference (Net) = -1.07, 95% CI [-2.12 to -0.02]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.580, t-test, 2 sided; Mean Difference (Net) = 0.30, 95% CI [-0.76 to 1.36]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.185, t-test, 2 sided; Mean Difference (Net) = -0.86, 95% CI [-2.14 to 0.41]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.438, t-test, 2 sided; Mean Difference (Net) = 0.51, 95% CI [-0.77 to 1.79]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.012, t-test, 2 sided; Mean Difference (Net) = 1.37, 95% CI [0.30 to 2.44]

34. Secondary Outcome: Change From Baseline to Week 13 Endpoint in the 36-item Short-Form Health Survey (SF36)- Mental Component Summary (MCS)
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.01 (1.11) | 0.57 (0.81) | -1.26 (0.82) | -0.45 (0.79)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.729, t-test, 2 sided; Mean Difference (Net) = 0.46, 95% CI [-2.16 to 3.08]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.352, t-test, 2 sided; Mean Difference (Net) = 1.02, 95% CI [-1.14 to 3.18]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.465, t-test, 2 sided; Mean Difference (Net) = -0.81, 95% CI [-3.00 to 1.37]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.677, t-test, 2 sided; Mean Difference (Net) = 0.56, 95% CI [-2.09 to 3.21]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.345, t-test, 2 sided; Mean Difference (Net) = -1.27, 95% CI [-3.92 to 1.38]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.102, t-test, 2 sided; Mean Difference (Net) = -1.84, 95% CI [-4.04 to 0.37]

35. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Physical Component Summary (PCS)
Description: as for outcome 34
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 6.07 (1.22) | 7.01 (0.88) | 7.85 (0.89) | 6.11 (0.86)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.977, t-test, 2 sided; Mean Difference (Net) = -0.04, 95% CI [-2.91 to 2.83]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.451, t-test, 2 sided; Mean Difference (Net) = 0.90, 95% CI [-1.44 to 3.24]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.150, t-test, 2 sided; Mean Difference (Net) = 1.74, 95% CI [-0.63 to 4.11]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.524, t-test, 2 sided; Mean Difference (Net) = 0.94, 95% CI [-1.96 to 3.83]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.230, t-test, 2 sided; Mean Difference (Net) = 1.78, 95% CI [-1.13 to 4.69]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.491, t-test, 2 sided; Mean Difference (Net) = 0.84, 95% CI [-1.55 to 3.23]

36. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Bodily Pain
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Bodily pain scores range from 2-11 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 1.51 (0.27) | 1.95 (0.20) | 2.11 (0.20) | 1.36 (0.19)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.645, t-test, 2 sided; Mean Difference (Net) = 0.15, 95% CI [-0.49 to 0.79]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.027, t-test, 2 sided; Mean Difference (Net) = 0.60, 95% CI [0.07 to 1.12]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Mean Difference (Net) = 0.75, 95% CI [0.22 to 1.29]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.180, t-test, 2 sided; Mean Difference (Net) = 0.44, 95% CI [-0.21 to 1.10]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.069, t-test, 2 sided; Mean Difference (Net) = 0.60, 95% CI [-0.05 to 1.25]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.564, t-test, 2 sided; Mean Difference (Net) = 0.16, 95% CI [-0.38 to 0.70]

37. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - General Health
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). General health scores range from 5-25(higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.70 (0.41) | 1.24 (0.30) | 0.81 (0.30) | 0.66 (0.29)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.929, t-test, 2 sided; Mean Difference (Net) = 0.04, 95% CI [-0.92 to 1.00]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.147, t-test, 2 sided; Mean Difference (Net) = 0.58, 95% CI [-0.21 to 1.36]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.700, t-test, 2 sided; Mean Difference (Net) = 0.16, 95% CI [-0.64 to 0.95]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.279, t-test, 2 sided; Mean Difference (Net) = 0.54, 95% CI [-0.44 to 1.51]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.822, t-test, 2 sided; Mean Difference (Net) = 0.11, 95% CI [-0.86 to 1.09]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.299, t-test, 2 sided; Mean Difference (Net) = -0.42, 95% CI [-1.22 to 0.38]

38. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Mental Health
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Mental health scores range from 5-30 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.21 (0.49) | 0.98 (0.36) | 0.46 (0.36) | 0.38 (0.35)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.766, t-test, 2 sided; Mean Difference (Net) = -0.18, 95% CI [-1.33 to 0.98]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.217, t-test, 2 sided; Mean Difference (Net) = 0.60, 95% CI [-0.35 to 1.55]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.880, t-test, 2 sided; Mean Difference (Net) = 0.07, 95% CI [-0.89 to 1.04]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.193, t-test, 2 sided; Mean Difference (Net) = 0.78, 95% CI [-0.39 to 1.94]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.675, t-test, 2 sided; Mean Difference (Net) = 0.25, 95% CI [-0.92 to 1.42]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.288, t-test, 2 sided; Mean Difference (Net) = -0.53, 95% CI [-1.50 to 0.45]

39. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Physical Functioning
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Physical functioning scores range from 10-30 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 1.80 (0.52) | 2.55 (0.38) | 3.11 (0.38) | 2.23 (0.37)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.501, t-test, 2 sided; Mean Difference (Net) = -0.42, 95% CI [-1.66 to 0.81]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.524, t-test, 2 sided; Mean Difference (Net) = 0.33, 95% CI [-0.69 to 1.35]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.089, t-test, 2 sided; Mean Difference (Net) = 0.89, 95% CI [-0.14 to 1.91]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.234, t-test, 2 sided; Mean Difference (Net) = 0.75, 95% CI [-0.49 to 2.00]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.040, t-test, 2 sided; Mean Difference (Net) = 1.31, 95% CI [0.06 to 2.56]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.289, t-test, 2 sided; Mean Difference (Net) = 0.56, 95% CI [-0.48 to 1.59]

40. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Role-Emotional
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Role-emotional scores range from 3-6 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.10 (0.12) | 0.19 (0.09) | 0.14 (0.09) | 0.08 (0.09)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.862, t-test, 2 sided; Mean Difference (Net) = 0.03, 95% CI [-0.27 to 0.32]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.368, t-test, 2 sided; Mean Difference (Net) = 0.11, 95% CI [-0.13 to 0.35]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.628, t-test, 2 sided; Mean Difference (Net) = 0.06, 95% CI [-0.18 to 0.31]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.573, t-test, 2 sided; Mean Difference (Net) = 0.09, 95% CI [-0.21 to 0.38]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.819, t-test, 2 sided; Mean Difference (Net) = 0.03, 95% CI [-0.26 to 0.33]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.687, t-test, 2 sided; Mean Difference (Net) = -0.05, 95% CI [-0.30 to 0.20]

41. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Role-Physical
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Role-physical scores range from 4-8 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.81 (0.21) | 0.80 (0.15) | 0.85 (0.15) | 0.80 (0.15)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.972, t-test, 2 sided; Mean Difference (Net) = 0.01, 95% CI [-0.48 to 0.50]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.990, t-test, 2 sided; Mean Difference (Net) = 0.00, 95% CI [-0.40 to 0.40]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.793, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI [-0.35 to 0.46]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.981, t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI [-0.50 to 0.49]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.857, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI [-0.45 to 0.54]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.805, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI [-0.36 to 0.46]

42. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Social Functioning
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Social functioning scores range from 2-10 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.75 (0.21) | 0.46 (0.16) | 0.38 (0.16) | 0.50 (0.15)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.340, t-test, 2 sided; Mean Difference (Net) = 0.24, 95% CI [-0.26 to 0.75]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.848, t-test, 2 sided; Mean Difference (Net) = -0.04, 95% CI [-0.45 to 0.37]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.573, t-test, 2 sided; Mean Difference (Net) = -0.12, 95% CI [-0.54 to 0.30]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.272, t-test, 2 sided; Mean Difference (Net) = -0.29, 95% CI [-0.79 to 0.22]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.161, t-test, 2 sided; Mean Difference (Net) = -0.36, 95% CI [-0.88 to 0.15]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.711, t-test, 2 sided; Mean Difference (Net) = -0.08, 95% CI [-0.50 to 0.34]

43. Secondary Outcome: Change From Baseline to Week 13 Endpoint in 36-Item Short-Form Health Survey (SF36) - Vitality
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). Vitality scores range from 4-24 (higher scores indicate better health status).
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 101 | 108
units on a scale | 0.69 (0.50) | 1.43 (0.36) | 0.44 (0.37) | 0.91 (0.35)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.713, t-test, 2 sided; Mean Difference (Net) = -0.22, 95% CI [-1.39 to 0.95]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.288, t-test, 2 sided; Mean Difference (Net) = 0.52, 95% CI [-0.44 to 1.49]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.351, t-test, 2 sided; Mean Difference (Net) = -0.46, 95% CI [-1.44 to 0.51]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.219, t-test, 2 sided; Mean Difference (Net) = 0.74, 95% CI [-0.44 to 1.93]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.686, t-test, 2 sided; Mean Difference (Net) = -0.24, 95% CI [-1.43 to 0.94]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.050, t-test, 2 sided; Mean Difference (Net) = -0.98, 95% CI [-1.97 to 0.00]

44. Secondary Outcome: Change From Baseline to Week 13 Endpoint in the Euro-Quality of Life Questionnaire - 5 Dimension - US Based Index Score
Description: The EuroQoL Questionnaire - 5 Dimension (EQ-5D) is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows patients to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 is generated for each domain. For each patient, the outcome rating on the 5 domains will be mapped to a single index through an algorithm. The index ranges between 0 and 1, with the higher score indicating a better health state perceived by the patient.
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 100 | 104
units on a scale | 0.04 (0.02) | 0.07 (0.01) | 0.08 (0.02) | 0.05 (0.01)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.663, t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI [-0.06 to 0.04]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.330, t-test, 2 sided; Mean Difference (Net) = 0.02, 95% CI [-0.02 to 0.06]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.143, t-test, 2 sided; Mean Difference (Net) = 0.03, 95% CI [-0.01 to 0.07]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.218, t-test, 2 sided; Mean Difference (Net) = 0.03, 95% CI [-0.02 to 0.08]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.100, t-test, 2 sided; Mean Difference (Net) = 0.04, 95% CI [-0.01 to 0.09]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.614, t-test, 2 sided; Mean Difference (Net) = 0.01, 95% CI [-0.03 to 0.05]

45. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Beck Depression Inventory-II Total Score
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 57 | 109 | 108 | 114
units on a scale | -1.24 (0.68) | -1.54 (0.50) | 0.37 (0.50) | -1.02 (0.49)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.786, t-test, 2 sided; Mean Difference (Net) = -0.22, 95% CI [-1.83 to 1.39]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.445, t-test, 2 sided; Mean Difference (Net) = -0.52, 95% CI [-1.85 to 0.81]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.043, t-test, 2 sided; Mean Difference (Net) = 1.39, 95% CI [0.04 to 2.74]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.721, t-test, 2 sided; Mean Difference (Net) = -0.30, 95% CI [-1.92 to 1.33]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.053, t-test, 2 sided; Mean Difference (Net) = 1.61, 95% CI [-0.02 to 3.24]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Mean Difference (Net) = 1.91, 95% CI [0.54 to 3.27]

46. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale
Description: A 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 54 | 102 | 100 | 106
units on a scale | -0.30 (0.36) | -0.81 (0.27) | -0.91 (0.27) | -0.68 (0.26)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.378, t-test, 2 sided; Mean Difference (Net) = 0.39, 95% CI [-0.48 to 1.25]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.723, t-test, 2 sided; Mean Difference (Net) = -0.13, 95% CI [-0.84 to 0.59]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.542, t-test, 2 sided; Mean Difference (Net) = -0.22, 95% CI [-0.95 to 0.50]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.245, t-test, 2 sided; Mean Difference (Net) = -0.52, 95% CI [-1.39 to 0.36]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.169, t-test, 2 sided; Mean Difference (Net) = -0.61, 95% CI [-1.48 to 0.26]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.796, t-test, 2 sided; Mean Difference (Net) = -0.10, 95% CI [-0.82 to 0.63]

47. Secondary Outcome: Adverse Events Reported as Reason for Discontinuation
Time Frame: Baseline to Week 13
Population: Number of all randomized patients.
Measure: Number; unit: participants
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 59 | 116 | 112 | 117
participants
  Patients Discontinued for Any Adverse Event | 9 | 17 | 27 | 10
  Insomnia | 1 | 1 | 3 | 0
  Nausea | 1 | 2 | 1 | 1
  Vomiting | 1 | 2 | 1 | 0
  Anxiety | 0 | 0 | 2 | 1
  Constipation | 1 | 1 | 1 | 0
  Diarrhoea | 0 | 1 | 0 | 1
  Dizziness | 0 | 0 | 1 | 1
  Dyspepsia | 0 | 1 | 0 | 1
  Erectile dysfunction | 0 | 2 | 0 | 0
  Hepatic enzyme increased | 0 | 1 | 1 | 0
  Somnolence | 1 | 0 | 1 | 0
  Abdominal pain | 1 | 0 | 0 | 0
  Abdominal pain upper | 0 | 0 | 1 | 0
  Apathy | 0 | 0 | 1 | 0
  Bursitis | 0 | 0 | 1 | 0
  Confusional state | 1 | 0 | 0 | 0
  Coordination abnormal | 0 | 0 | 0 | 1
  Decreased appetite | 0 | 0 | 1 | 0
  Disturbance in attention | 0 | 1 | 0 | 0
  Dysphoria | 1 | 0 | 0 | 0
  Ejaculation disorder | 0 | 0 | 1 | 0
  Fatigue | 0 | 0 | 1 | 0
  Gastroenteritis | 0 | 0 | 1 | 0
  Glaucoma | 0 | 0 | 0 | 1
  Headache | 0 | 0 | 0 | 1
  Hepatitis | 0 | 1 | 0 | 0
  Hot flush | 0 | 1 | 0 | 0
  Hyperhidrosis | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 1 | 0
  Irritability | 1 | 0 | 0 | 0
  Lethargy | 0 | 0 | 1 | 0
  Loss of libido | 0 | 0 | 1 | 0
  Muscular weakness | 0 | 1 | 0 | 0
  Myocardial infarction | 0 | 0 | 1 | 0
  Palpitations | 0 | 1 | 0 | 0
  Peritonsillar abscess | 0 | 0 | 0 | 1
  Pregnancy | 0 | 0 | 0 | 1
  Rash | 0 | 1 | 0 | 0
  Restless legs syndrome | 0 | 0 | 1 | 0
  Sedation | 0 | 0 | 1 | 0
  Testicular pain | 0 | 0 | 1 | 0
  Trismus | 0 | 0 | 1 | 0

48. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessments - Alkaline Phosphatase
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 107 | 104 | 113
Units/Liter | -1.19 (11.19) | 3.27 (14.17) | 1.11 (12.37) | -1.43 (7.61)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.015, t-test, 2 sided
Statistical Analysis 3: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.015, t-test, 2 sided

49. Secondary Outcome: Change From Baseline to 13 Week Endpoint in Laboratory Assessments - Alanine Transaminase
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 106 | 104 | 112
Units/Liter | -1.39 (10.91) | 0.25 (21.53) | 2.20 (12.45) | -0.06 (9.48)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.039, t-test, 2 sided

50. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Bicarbonate, HCO3
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 57 | 106 | 104 | 112
millimole/Liter | 1.04 (3.29) | 1.18 (3.60) | 1.72 (2.93) | 1.35 (3.09)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.048, t-test, 2 sided

51. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Bilirubin, Direct
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 105 | 102 | 112
micromole/Liter | -0.29 (0.68) | -0.13 (0.82) | -0.13 (0.74) | 0.07 (0.82)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.015, t-test, 2 sided
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.046, t-test, 2 sided

52. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Bilirubin, Total
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 57 | 106 | 104 | 113
micromole/Liter | -1.05 (2.56) | -0.23 (3.50) | -0.58 (2.57) | 0.18 (3.15)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.039, t-test, 2 sided

53. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Chloride
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 107 | 104 | 114
millimole/Liter | -0.22 (2.44) | -0.54 (2.81) | -0.99 (2.55) | -0.47 (2.48)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.042, t-test, 2 sided

54. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Cholesterol
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 107 | 104 | 114
millimole/Liter | -0.04 (0.74) | -0.09 (0.70) | 0.01 (0.88) | -0.22 (0.62)
Statistical Analysis 1: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

55. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Creatinine
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 107 | 104 | 114
micromole/Liter | -11.43 (89.68) | -0.66 (8.96) | 1.34 (9.91) | 2.02 (10.36)
Statistical Analysis 1: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.031, t-test, 2 sided

56. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Potassium
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 56 | 107 | 104 | 113
millimole/Liter | -0.02 (0.41) | 0.00 (0.42) | 0.06 (0.44) | -0.08 (0.42)
Statistical Analysis 1: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.030, t-test, 2 sided

57. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Laboratory Assessment - Uric Acid
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 107 | 104 | 114
micromole/Liter | -9.48 (45.82) | -11.08 (49.35) | -11.31 (50.54) | 8.20 (37.89)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

58. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Vital Signs - Pulse Rate
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 110 | 108 | 114
beats per minute | -1.10 (1.21) | 2.79 (0.89) | 1.90 (0.90) | 0.29 (0.87)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.348, t-test, 2 sided; Mean Difference (Net) = -1.38, 95% CI [-4.28 to 1.51]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.040, t-test, 2 sided; Mean Difference (Net) = 2.50, 95% CI [0.11 to 4.89]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.191, t-test, 2 sided; Mean Difference (Net) = 1.61, 95% CI [-0.81 to 4.03]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Mean Difference (Net) = 3.89, 95% CI [0.97 to 6.80]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.044, t-test, 2 sided; Mean Difference (Net) = 3.00, 95% CI [0.08 to 5.91]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.473, t-test, 2 sided; Mean Difference (Net) = -0.89, 95% CI [-3.33 to 1.55]

59. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Vital Signs - Systolic Blood Pressure
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 110 | 108 | 114
mm Hg | -0.64 (1.68) | -1.18 (1.24) | 1.00 (1.25) | -1.04 (1.21)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.846, t-test, 2 sided; Mean Difference (Net) = 0.40, 95% CI [-3.61 to 4.40]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.934, t-test, 2 sided; Mean Difference (Net) = -0.14, 95% CI [-3.45 to 3.17]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.234, t-test, 2 sided; Mean Difference (Net) = 2.03, 95% CI [-1.32 to 5.39]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.794, t-test, 2 sided; Mean Difference (Net) = -0.54, 95% CI [-4.58 to 3.50]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.426, t-test, 2 sided; Mean Difference (Net) = 1.64, 95% CI [-2.40 to 5.67]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.207, t-test, 2 sided; Mean Difference (Net) = 2.17, 95% CI [-1.21 to 5.55]

60. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Vital Signs - Diastolic Blood Pressure
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 110 | 108 | 114
mm Hg | -0.51 (1.14) | -0.79 (0.84) | 2.94 (0.85) | -0.68 (0.82)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.901, t-test, 2 sided; Mean Difference (Net) = 0.17, 95% CI [-2.54 to 2.89]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.926, t-test, 2 sided; Mean Difference (Net) = -0.11, 95% CI [-2.35 to 2.14]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Net) = 3.62, 95% CI [1.35 to 5.90]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.841, t-test, 2 sided; Mean Difference (Net) = -0.28, 95% CI [-3.02 to 2.46]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.014, t-test, 2 sided; Mean Difference (Net) = 3.45, 95% CI [0.71 to 6.19]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Net) = 3.73, 95% CI [1.44 to 6.02]

61. Secondary Outcome: Change From Baseline to Week 13 Endpoint in Vital Signs - Weight
Time Frame: Baseline, Week 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Number analyzed (Participants) | 58 | 110 | 108 | 114
kilograms | -0.59 (0.30) | -0.35 (0.22) | -0.72 (0.22) | 0.10 (0.22)
Statistical Analysis 1: Comparison: Duloxetine 20 mg vs Placebo; Test type: Superiority or Other; p = 0.057, t-test, 2 sided; Mean Difference (Net) = -0.70, 95% CI [-1.41 to 0.02]
Statistical Analysis 2: Comparison: Duloxetine 60 mg vs Placebo; Test type: Superiority or Other; p = 0.128, t-test, 2 sided; Mean Difference (Net) = -0.46, 95% CI [-1.05 to 0.13]
Statistical Analysis 3: Comparison: Duloxetine 120 mg vs Placebo; Test type: Superiority or Other; p = 0.007, t-test, 2 sided; Mean Difference (Net) = -0.82, 95% CI [-1.42 to -0.22]
Statistical Analysis 4: Comparison: Duloxetine 20 mg vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.518, t-test, 2 sided; Mean Difference (Net) = 0.24, 95% CI [-0.48 to 0.96]
Statistical Analysis 5: Comparison: Duloxetine 20 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.734, t-test, 2 sided; Mean Difference (Net) = -0.12, 95% CI [-0.85 to 0.60]
Statistical Analysis 6: Comparison: Duloxetine 60 mg vs Duloxetine 120 mg; Test type: Superiority or Other; p = 0.239, t-test, 2 sided; Mean Difference (Net) = -0.36, 95% CI [-0.97 to 0.24]

ADVERSE EVENTS:
Arm/Group | Duloxetine 20 mg | Duloxetine 60 mg | Duloxetine 120 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/116 | 3/112 | 3/117
Other Adverse Events (participants affected / at risk) | 39/59 | 78/116 | 80/112 | 69/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 20 mg (N=59) | Duloxetine 60 mg (N=116) | Duloxetine 120 mg (N=112) | Placebo (N=117)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 20 mg (N=59) | Duloxetine 60 mg (N=116) | Duloxetine 120 mg (N=112) | Placebo (N=117)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 10 (10) | 14 (14) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 10 (12) | 7 (8) | 4 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 12 (13) | 12 (12) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (12) | 24 (24) | 14 (14) | 4 (6)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 7 (7) | 10 (10) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Irritability (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Therapeutic response unexpected (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 6 (6) | 5 (5) | 5 (5)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Pharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurological examination abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 9 (9) | 9 (9) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 12 (15) | 10 (17) | 4 (4)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 5 (5) | 14 (14) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Anorgasmia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 10 (11) | 21 (22) | 3 (3)
Libido decreased (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejaculation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days